CLINICAL TRIAL: NCT06047769
Title: Effects of Board Games on Balance in Association With Cognition in Community-Dwelling Elderly.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: REC01539 Muhammad Ammar
Record Dates: First submitted 2023-09-14; First posted 2023-09-21 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2024-05

CONDITIONS: Geriatric Population

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional Group (Experimental): Participants will receive cognitive training in board games including Ludo, Chutes & Ladder and Chess with both single and multiplayer modes. After 1 week of training, participants will receive intervention of 1 hour per day, three days a week for 8 weeks completing a total of 1440 minutes. With this technique, we will target the cognitive process of information processing, speed and executive function of the patient.
  Interventions: Other: Board Games
- Control group (No Intervention): Participants will receive no intervention and will be observed for 8 weeks.

INTERVENTIONS:
Other: Board Games — Participants will receive cognitive training in board games including Ludo, Chutes & Ladder and Chess with both single and multiplayer modes. After 1 week of training, participants will receive intervention of 1 hour per day, three days a week for 8 weeks completing a total of 1440 minutes. With this technique, we will target the cognitive process of information processing, speed and executive function of the patient.
  Arms: Interventional Group

SUMMARY:
As age progress incidence of fall increases. Cognitively impaired patients have poor balance and they are more prone to falls. Balance and cognitive functions are co-related in middle-aged and community-dwelling elderly. In fact age-related cognitive decline as the brain ages it has exceptional neuroplasticity. To maintain balance and prevent falls various cognitive processes are required. Board games can be used as tools for cognitive training as they have the means to restore and form motor skills, cognitive functioning, and logical and spatial thinking. Cognitive training using simple games might improve the elements of balance and gait, and prevent falls.

DETAILED DESCRIPTION:
In fact age-related cognitive decline, as the brain ages, it has exceptional neuroplasticity. This can be achieved by cognitive training which consists of domain-specific task completion or exercises to promote neurogenesis in that domain. Cognitive training is an approach towards enhancing neural plasticity by focusing on and training cognitive domains for balance improvement. Board games can be used as tools for cognitive training as they have the means to restore and form motor skills, cognitive functioning, and logical and spatial thinking. A board game is a generic term for a game played by placing, moving or removing pieces on a board and that utilizes a game format in which pieces are moved in particular ways on a board marked with a pattern. As a tool, board games can improve comprehension and cognitive functioning among participants.

As per a study, computer-based cognitive training by simple games such as Road Tour, Jewel Diver, and Sweep Seeker improved visuospatial memory, speed of processing and inhibition which in turn improved balance and gait, and prevented falls in community-dwelling elderly but as per the author's access, there's lack of standardization in terms of types of cognitive training program intended to improve balance in the elderly population by using simple board games. Hence, the author established the research question of whether is this technique effective in the elderly population in terms of its effects on cognition and balance to prevent falls. This study will provide insight to the clinician on whether board games-based cognitive training improves balance and prevents fall risk in the elderly population.

ELIGIBILITY:
Inclusion Criteria:

* Males and Female participants aged 60 years or older.
* Score of 26 or more on the Mini-Mental State Examination (MMSE)
* At least one self-reported fall within the last 2 years or (BBS) score less than 52 and more than 41.
* Subjects who are willing to commit to the time commitments required by the program.

Exclusion Criteria:

* Those who will not meet the inclusion criteria.
* Presence of any physical limitation that may limit hand movement.
* Presence of a severe walking or balance impairment For Example; (Amputation, or Fracture at that time.)
* Self-reported presence of vertigo
* Any visual disease
* Currently using psychotropic medications.
* Presence of any neurological disorder

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2023-09-22 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-01-30 (Actual)

PRIMARY OUTCOMES:
Berg Balance Scale (BBS) | Baseline
  A testing tool with high validity ( 0.93) and reliability (0.98) was used to measure balance in the elderly. The Berg Balance Scale (BBS) is a valid tool. The total score for the BBS is 56 and a higher score means good balance. It will be measured at baseline, 4th week and 8th week.
Berg Balance Scale (BBS) | After 4 weeks
  A testing tool with high validity ( 0.93) and reliability (0.98) was used to measure balance in the elderly. The Berg Balance Scale (BBS) is a valid tool. The total score for the BBS is 56 and a higher score means good balance. It will be measured at baseline, 4th week and 8th week.
Berg Balance Scale (BBS) | After 8 weeks
  A testing tool with high validity ( 0.93) and reliability (0.98) was used to measure balance in the elderly. The Berg Balance Scale (BBS) is a valid tool. The total score for the BBS is 56 and a higher score means good balance. It will be measured at baseline, 4th week and 8th week.
Mini-Mental State Exam (MMSE) | Baseline
  A set of 11 questions that doctors and other healthcare professionals commonly use to check for cognitive impairment (problems with thinking, communication, understanding and memory) with reliability of (0.98) and reliability (0.77). The Mini-Mental State Exam (MMSE) is a valid tool. It will be measured at baseline, 4th week and 8th week. The total score for the MMSE is 30 and a higher score means good cognition.
Mini-Mental State Exam (MMSE) | After 4 weeks
  A set of 11 questions that doctors and other healthcare professionals commonly use to check for cognitive impairment (problems with thinking, communication, understanding and memory) with reliability of (0.98) and reliability (0.77). The Mini-Mental State Exam (MMSE) is a valid tool. It will be measured at baseline, 4th week and 8th week. The total score for the MMSE is 30 and a higher score means good cognition.
Mini-Mental State Exam (MMSE) | After 8 weeks
  A set of 11 questions that doctors and other healthcare professionals commonly use to check for cognitive impairment (problems with thinking, communication, understanding and memory) with reliability of (0.98) and reliability (0.77). The Mini-Mental State Exam (MMSE) is a valid tool. It will be measured at baseline, 4th week and 8th week. The total score for the MMSE is 30 and a higher score means good cognition.

SECONDARY OUTCOMES:
Dynamic Gait Index (DGI) | Baseline
  A clinical tool to assess gait, balance and fall risk with reliability of (0.98). The Dynamic Gait Index (DGI) is a valid tool. It will be measured at baseline, 4th week and 8th week. The total possible score is 24. A lower score indicates greater impairment or a higher risk of falls.
Dynamic Gait Index (DGI) | After 4 weeks
  A clinical tool to assess gait, balance and fall risk with reliability of (0.98). The Dynamic Gait Index (DGI) is a valid tool. It will be measured at baseline, 4th week and 8th week. The total possible score is 24. A lower score indicates greater impairment or a higher risk of falls.
Dynamic Gait Index (DGI) | After 8 weeks
  A clinical tool to assess gait, balance and fall risk with reliability of (0.98). The Dynamic Gait Index (DGI) is a valid tool. It will be measured at baseline, 4th week and 8th week. The total possible score is 24. A lower score indicates greater impairment or a higher risk of falls.
Timed Up & Go test (TUG) | Baseline
  It is a quick and widely used clinical performance-based measure of lower extremity function, mobility and fall risk with a specificity of 0.70 sensitivity of 0.57(17) and reliability of (0.98). The Timed Up & Go test (TUG) test is a valid tool. The TUG is timed. The score is the time (in seconds) it takes the person to complete the task, starting from the command "Go" and stopping when the person is seated back in the chair. Times greater than 13.5 seconds are often associated with a higher risk of falls. It will be measured at baseline, 4th week and 8th week.
Timed Up & Go test (TUG) | After 4 weeks
  It is a quick and widely used clinical performance-based measure of lower extremity function, mobility and fall risk with a specificity of 0.70 sensitivity of 0.57(17) and reliability of (0.98). The Timed Up & Go test (TUG) test is a valid tool. The TUG is timed. The score is the time (in seconds) it takes the person to complete the task, starting from the command "Go" and stopping when the person is seated back in the chair. Times greater than 13.5 seconds are often associated with a higher risk of falls. It will be measured at baseline, 4th week and 8th week.
Timed Up & Go test (TUG) | After 8 weeks
  It is a quick and widely used clinical performance-based measure of lower extremity function, mobility and fall risk with a specificity of 0.70 sensitivity of 0.57(17) and reliability of (0.98). The Timed Up & Go test (TUG) test is a valid tool. The TUG is timed. The score is the time (in seconds) it takes the person to complete the task, starting from the command "Go" and stopping when the person is seated back in the chair. Times greater than 13.5 seconds are often associated with a higher risk of falls. It will be measured at baseline, 4th week and 8th week.

CONTACTS AND LOCATIONS:
Overall Officials: Imran Amjad, PhD, Principal Investigator — Riphah International University
Locations (1):
- ABID Hospital, Islamabad, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Smith-Ray RL, Hughes SL, Prohaska TR, Little DM, Jurivich DA, Hedeker D. Impact of Cognitive Training on Balance and Gait in Older Adults. J Gerontol B Psychol Sci Soc Sci. 2015 May;70(3):357-66. doi: 10.1093/geronb/gbt097. Epub 2013 Nov 5. PMID 24192586
- [Background] Smith-Ray RL, Makowski-Woidan B, Hughes SL. A randomized trial to measure the impact of a community-based cognitive training intervention on balance and gait in cognitively intact Black older adults. Health Educ Behav. 2014 Oct;41(1 Suppl):62S-9S. doi: 10.1177/1090198114537068. PMID 25274713
- [Background] Willis SL, Tennstedt SL, Marsiske M, Ball K, Elias J, Koepke KM, Morris JN, Rebok GW, Unverzagt FW, Stoddard AM, Wright E; ACTIVE Study Group. Long-term effects of cognitive training on everyday functional outcomes in older adults. JAMA. 2006 Dec 20;296(23):2805-14. doi: 10.1001/jama.296.23.2805. PMID 17179457
- [Background] Noda S, Shirotsuki K, Nakao M. The effectiveness of intervention with board games: a systematic review. Biopsychosoc Med. 2019 Oct 21;13:22. doi: 10.1186/s13030-019-0164-1. eCollection 2019. PMID 31641371
- [Background] Smith GE, Housen P, Yaffe K, Ruff R, Kennison RF, Mahncke HW, Zelinski EM. A cognitive training program based on principles of brain plasticity: results from the Improvement in Memory with Plasticity-based Adaptive Cognitive Training (IMPACT) study. J Am Geriatr Soc. 2009 Apr;57(4):594-603. doi: 10.1111/j.1532-5415.2008.02167.x. Epub 2009 Feb 9. PMID 19220558